CLINICAL TRIAL: NCT06954909
Title: The Impact of Self-assessment on Wildland Firefighter and Surrogate Population Hydration
Brief Title: The Impact of Self-assessment on Hydration
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Floris Wardenaar, Assistant Professor in Nutrition, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EMW-2022- FP-00082; EMW-2022- FP-00082 (Other Grant/Funding Number: DHS: Federal Emergency Management Agency (FEMA))
Record Dates: First submitted 2025-04-17; First posted 2025-05-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hydration Status
Keywords: Urine osmolality; Urine specific gravity; Labelled water (D20); Deuterium; Education; Self-assessment; Tactical operators; Firefighters; Women; Men; Healthy subjects
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Intervention Model Description: Allocation to intervention (INT) or control (CON) depends on the total number of participants at different locations that will be eligible. The investigators will try to match participants based on their sex, age and bodyweight, and then randomly assign these matched participants to the intervention or control group. The control group participants will be offered to follow the education session after data collection has been finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydration education and hydration self-assessment (Experimental): Participants will participate in a 25-minute hydration education session that also includes instruction about how the use the hydration self-assessment worksheets and materials.
  Interventions: Behavioral: Hydration education and self-assessment
- No Hydration education and hydration self-assessment (business as usual) (No Intervention): Participants do not participate in any education or self-assessment, other than applying their normal hydration strategies.

INTERVENTIONS:
Behavioral: Hydration education and self-assessment — Hydration education is a 25-minute session based on the theory of planned behavior, including the instructions how to use a worksheet for hydration self-assessment and materials.
  Arms: Hydration education and hydration self-assessment

SUMMARY:
The studies objective is to assess the efficacy of hydration education and the use of a self-assessment worksheet vs. a no-intervention control on improving fluid intake and hydration status in underhydrated wildland firefighters (WLFFs) and their surrogates.

Part I allows to understand hydration status of the participants (screening phase), Part II confirms if participants indeed are deemed to be low fluid consumers, and Part III of this research is a clinical trial that will focus on the optimization of hydration by improving fluid intake (and as a result lowering urine concentration) allowing participants theoretically to improve exercise performance (acute) and optimize health on the long term.

DETAILED DESCRIPTION:
Enrollment will take place until enough people have been screened and be eligible to be enrolled in PART III of the study.

Aside from allowing the investigators to better understand the hydration status of participants in PART I, this part will help to determine potentially eligible participants that can be confirmed through PART II by collecting again a urine sample, and if again concentrated urine is confirmed the research team will take a 5 mL venous blood draw performed by a trained phlebotomist to confirm elevated a copeptin level. These confirmed participants can then be enrolled in PART III of the study when eligible.

PART I includes all participants:

Two urine samples and questionnaire at one day. Expected duration of 2-3 minutes per urine sample and 2-3 minutes for the participant demographics questionnaire which will also be used as a screener to identify eligibility for PART II and III.

PART II includes a smaller sample:

Collection of a urine sample and a blood sample at one follow up day for the duration of 10 minutes.

PART III, the intervention study (being a clinical trial):

Includes n=38 participants, that will invest a maximum of 2 hours and 15 minutes as part of the data collection over a period of 6 days, which includes:

* Education session (pre: INT, or post: CON) of 25 minutes.
* Consuming labelled water and providing a urine sample and bodyweight the day before the start of the study, 10-15 minutes.
* Participate in the study for 6 days (during normal work days) and bodyweight will be measured at day 2, 4 and 6 of the study, during all study days both INT and CON will provide a morning urine sample (and if possible an afternoon/evening sample after work), and during each days sensors will be attached to participants upper arm and gear, 5 minutes per day, 25-30 minutes total.
* The intervention group will track its use of the tools we have provided them with, while the other group will not perform any additional self-assessments during the study period, 10 minutes per day 25-50 minutes total.
* Final hydration strategy questionnaire for INT and CON, 5-10 minutes.

Allocation to INT or CON depends on the total number of participants at different locations that will be eligible. The investigators will try to match participants based on their sex, age and bodyweight, and then randomly assign these matched participants to the intervention or placebo.

ELIGIBILITY:
The study plans to include firefighters from the Tonto National Forest and the broader Phoenix Valley area, and if needed, other active populations that are similarly active to WLFFs. Participants with high urine concentration (≥1.020 USG) for both samples collected during Part I (screening phase), may be invited to provide an additional urine sample and a blood sample for copeptin analysis during a follow up day (Part II). Participants with elevated USG and copeptin are eligible to participate in the study.

Inclusion for PART I is that participants are part of a by the research selected wildland firefighter population (or surrogate population), no further exclusion criteria are followed for PART I. For Part II and Part III the following criteria apply:

Inclusion Criteria:

* Age 18-65 years
* Identifying as male, female or other

Exclusion Criteria:

* Thyroid medication
* Bariatric surgery
* Cardiovascular disease
* Renal disease
* Hepatic disease
* Bodyweight <110 lbs.
* Any injury that would not allow physical performance or activity
* Pregnant or lactating
* Diuretics
* Non-stable self-reported body weight for the last month (<10 lbs. fluctuation)

Investigators will not exclude participants reporting the use of dietary supplements as there is no evidence that the accuracy of self-assessment (specifically the accuracy of urine color assessment) to determine a low vs. high urine concentration is influenced by dietary supplement use, but participants will be questioned about their supplement, electrolyte and sport drink use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Fluid turnover | Over a period of 4 days, in two 48-hour segments.
  Fluid turnover based on D2O analysis
Urine concentration | Afternoon sample day 1, morning sample day 2/4/6
  Urine concentration (osmolality).

SECONDARY OUTCOMES:
Urine concentration | Afternoon sample day 1, morning (and potential afternoon) samples day 1/2/3/4/5/6.
  Urine concentration (USG ) for morning and when available afternoon/evening samples.
Activity | Throughout the study during working hours, which may vary between 8-16 hours per working day.
  Activity pattern using an activity tracker attached to the upper arm to allow comparing activity between INT and CON.
Hydration strategy | Day 6 of the data collection, covering the hydration strategy during the study period.
  Retrospective hydration strategy (questionnaire) of INT and CON.
Heat stress | Throughout the study during working hours, which may vary between 8-16 hours per working day.
  Direct experienced environmental heat, measured by a heat sensor mounted on helmet or gear.
INT: Self-reported hydration measures | Study days 2/3/4/5/6.
  Self-reported hydration measures in INT only (daily fluid intake in mL).
INT: Self-reported hydration measures | Study days 2/3/4/5/6.
  Self-reported hydration measures in INT only (urine frequency, number of voids per 24-hour).
INT: Self-reported hydration measures | Study days 2/3/4/5/6.
  Self-reported hydration measures in INT only (first morning urine volume in mL).
INT: Self-reported hydration measures | Study days 2/3/4/5/6.
  Self-reported hydration measures in INT only (urine color, assessed on a scale from 1-7 ranging from light to dark).

OTHER OUTCOMES:
Demographics | Measured at the start of the study during Part I (screening phase).
  Personal demographics, such as age, sex, race, ethnicity, work location, work status, short medical history, use of medication, use of dietary supplements, electrolyte and sports drinks, alcohol and tobacco use (questionnaire)
Environmental conditions | Throughout the study during working hours, which may vary between 8-16 hours per working day.
  Environmental measurements using a local weather station to be able to report ambient temperature in degrees Celsius.
Environmental conditions | Throughout the study during working hours, which may vary between 8-16 hours per working day.
  Environmental measurements using a local weather station to be able to report relative humidity (%).
Environmental conditions | Throughout the study during working hours, which may vary between 8-16 hours per working day.
  Environmental measurements using a local weather station to be able to report solar radiation in watts per square meter (W/m2 = Wm-2).

CONTACTS AND LOCATIONS:
Locations (1):
- ASU Health Futures Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wardenaar FC, Thompsett D, Vento KA, Bacalzo D. A lavatory urine color (LUC) chart method can identify hypohydration in a physically active population. Eur J Nutr. 2021 Aug;60(5):2795-2805. doi: 10.1007/s00394-020-02460-5. Epub 2021 Jan 8. PMID 33416980